CLINICAL TRIAL: NCT06418321
Title: Early Identification of Age-related Hearing Impairment
Status: Completed | Type: Observational
Sponsor: Aalto University (Other)
Collaborators: Business Finland (Other); Helsinki University Central Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 535/2024
Record Dates: First submitted 2024-04-15; First posted 2024-05-17 (Actual); Last update posted 2025-02-20 (Actual); Status verified 2025-02

CONDITIONS: Hearing Loss, Age-Related
MeSH Terms: conditions — Presbycusis | interventions — Sleep, REM

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Participant group 1: HUS Helsinki University Hospital: Participants are tested with the investigational device and the gold-standard device.
  Interventions: Device: Investigational device; Other: Audiometer; Device: Otomicroscopy; Other: REM (Real Ear Measurements)
- Participant group 2: Aalto University: Participants are tested with the investigational device.
  Interventions: Device: Investigational device

INTERVENTIONS:
Device: Investigational device — The participants' hearing status will be evaluated using the investigational device.
Other: Audiometer — Participants' hearing thresholds are tested with an audiogram.
  Groups: Participant group 1: HUS Helsinki University Hospital
Device: Otomicroscopy — The status of the participants' ear canals and tympanic membranes are checked.
  Groups: Participant group 1: HUS Helsinki University Hospital
Other: REM (Real Ear Measurements) — The acoustic properties of the participants' ears will be measured during the interventions.
  Groups: Participant group 1: HUS Helsinki University Hospital

SUMMARY:
The need for future hearing rehabilitation is enormous. World Health Organization (WHO 2021) has estimated that by 2050, 2.5 billion people will have some degree of hearing loss, and 1/4 of them will require hearing rehabilitation. Currently, healthcare systems and processes are already overwhelmed and not adequately equipped to screen and diagnose this rapidly growing population suffering from hearing impairment. This study aims to investigate if the diagnostics of age-related hearing loss can be accelerated by involving patients in the hearing assessment process.

DETAILED DESCRIPTION:
The investigational device used in the study is part of the Otoscreen hearing screening system that is developed by Aalto University.

The investigational device consists of the following parts:

* Digital otoscope
* User interface control unit.

The investigational device is designed to record high-quality images and videos of the eardrum and ear canal and guide users through a hearing screening test while collecting data from questionnaires, digital otoscopy, and audiometry.

The investigational device is used together with a CE-marked audiometer that is intended for hearing screening testing.

ELIGIBILITY:
Inclusion Criteria:

• Must be able to understand Finnish or Swedish

Exclusion Criteria:

• Clinical diagnosis of hearing loss

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy volunteers
Sampling Method: Probability Sample
Enrollment: 49 (Actual)
Dates: Start 2024-04-04 (Actual); Primary Completion 2025-02-12 (Actual); Study Completion 2025-02-12 (Actual)

PRIMARY OUTCOMES:
Comparison between investigational device and gold-standard device (otomicroscope) findings. | From digital otoscopy to the interpretation of pictures (up to six months).
  The investigators compare scored views to the outer ear canal and tympanic membrane.
Comparison between the automated hearing screening self-test result and the gold-standard hearing test result performed with clinical Audiometer by an Audiologist. | From hearing tests to the comparison (up to six months).
  The investigators compare pure tone averages.

SECONDARY OUTCOMES:
Participant group 2: The usability of the investigational device. | From study appointment to the analysis of the results (up to six months).
  The usability of the investigational device will be assessed using a usability testing protocol. It includes subjective feedback from participants through interviews, questionnaires, and observation of device use. The usability will be assessed using the AttrakDiff method, a standardized questionnaire designed to measure the user's perception of a product's attractiveness, pragmatism, and overall appeal. This method provides insights into both the pragmatic and hedonic aspects of usability. AttrakDiff consists of multiple items scored on a semantic differential scale that consists of seven-step items whose poles are opposite adjectives (e.g. "confusing - clear", "unusual - ordinary", "good - bad"). Each set of adjective items is ordered into a scale of intensity.
  Usability testing will be conducted iteratively with the first group of participants (N=20), followed by modifications based on feedback. This iterative process will continue until no negative feedback is received.
Participant group 1: REM measurements. | From REM measurements to the analysis of the results (up to six months).
  If there is a difference between the automated hearing screening self-test result and the gold-standard hearing test result performed with clinical Audiometer, the investigators will look for the REM results if there is an explanation for the difference at the individual level.

CONTACTS AND LOCATIONS:
Overall Officials: Jouni Partanen, Prof., Principal Investigator — Aalto University
Locations (2):
- Finland (2):
  - Aalto University, Espoo
  - HUS Head and Neck Center, Helsinki